CLINICAL TRIAL: NCT00267644
Title: Ultrasound of the Inferior Vena Cava (IVC) and Dehydration Status in Pediatric Emergency Patients
Status: Completed | Type: Observational
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Manager, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Other Study IDs: 05-09-VA03
Record Dates: First submitted 2005-12-19; First posted 2005-12-21 (Estimated); Results first posted 2013-07-03 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-04

CONDITIONS: Dehydration
Keywords: Children, dehydration, Ultrasound
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Hydrated patients: Group 1 (n=63) were pediatric patiens that wer hydrated.
- Dehydrated Group: Group 2 (n=13) were pediatric patients that were dehydrated.

SUMMARY:
Objective: Although approximately 9% of patients presenting to a Pediatric Emergency Department (ED) are dehydrated, there is no reliable method to measure objectively the degree of intravascular dehydration. Respiratory changes in Inferior Vena Cava (IVC) diameter have been shown to predict volume status in adults. Previous research has demonstrated correlation between IVC diameter and volume status in children undergoing hemodialysis. Other studies have shown that IVC diameter in children can be sonographically measured rapidly and accurately by ED physicians. If we can establish that IVC diameter predicts volume status in dehydrated children, this tool could assist the ED physician in rapid diagnosis and prompt resuscitation without the need to wait for blood or urine tests. In this study we use the "dehydrated patient" as a model for hypovolemia, with the idea that the data could ultimately be used in the setting of any hypovolemic state. We aim to evaluate whether ultrasound of the pediatric IVC can be used to reliably assess volume status.

Methods: This is a prospective cohort study. Pediatric ED patients ranging in age from 1 to 41 months were assessed by a Pediatric emergency physician and stratified as either clinically euvolemic or hypovolemic. After consent was obtained, one of three Emergency Medicine Residents performed trans-abdominal sonographic measurements of the IVC diameter. Measurements of the IVC diameter just caudal to the insertion of the hepatic veins were obtained in a longitudinal orientation.

DETAILED DESCRIPTION:
Ultrasound is considered a routine procedure in the ED. In MMC all ultrasound done by ED staff is documented, however patients are not billed for it. All the ultrasound images for this study will have to be approved by Dr. Marshall prior to inclusion into the study.

For the purposes of this study, trans-abdominal ultrasonographic measurements of the Inferior Vena Cava (IVC) will be taken in patients suspected of being Dehydrated. The Triage Nurse will be the person who would identify acutely dehydrated patient. Once a potential candidate is identified The Attending physician in the pediatric ED will be notified. If a sonographer is available in the ED at the time and he/she is free/willing to perform the sonogram only then will the attending physician will notify and consent the patient.

The first phase of the study will concentrate on establishing the correlation between collapsed IVC and level of dehydration. During the first part of the study, ultrasonography will be performed once prior to hydration.

During this phase we will also perform sonograms on a control group. The Control Group will consist of children aged 1 month to 3 years age who we do not suspect of being dehydrated based on initial evaluation and presenting complaints.

During the second phase of the study we will measure the change in IVC diameter with fluid resuscitation. During this time, additional ultrasonography will be performed after adequate fluid resuscitation.

Return Visit: For the patient that qualify for a return visit for a weight check, upon arrival to the ED, will bypass registration and report to the triage nurse and identify themselves, where they will be weighed and then promptly sent home.

Who needs a return visit? Any patient who is not admitted or does not have a recent weight available (at the PMD's office) prior to the onset of the current condition will qualify for a return visit. The patients who has a recent weight taken at the PMD's office will be requested to sign the hospitals standard consent for transfer of the data via fax from the PMD's office.

ELIGIBILITY:
Inclusion Criteria:Any patient 1-month to 36 months of age presenting to the ED with a History or vomiting, Diarrhea or decreased PO intake in which the Attending physician is concerned about Dehydration (cases) and patients in the same age group who are not suspected of dehydration (controls).

-

Exclusion Criteria:

a. Presentation to the ED is more than 5 days from onset of symptoms. b. Upon initial evaluation patient who are thought to need immediate resuscitation will be excluded for the study.

-

Ages: 1 Month to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Any ED patient 1-month to 41 months of age presenting to the ED with a History or vomiting, Diarrhea or decreased PO intake
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2005-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hashibul Hannan, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the Pediatric ED from
Pre-assignment Details: NO patient was excluded from the trial
Groups:
- Cases: Dehydrated Pediatric Patients
- Controls: Hydrated Pediatric Patients
Period: Overall Study
Arm/Group | Cases | Controls
Started | 13 | 63
Completed | 13 | 63
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cases | Controls | Total
Number analyzed (Participants) | 13 | 63 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 63 | 76
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 1.6 (.83) | 1.2 (.41) | 1.5 (.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 36 | 40
  Male | 9 | 27 | 36
Region of Enrollment [Number; unit: participants]
  United States | 13 | 63 | 76

OUTCOME MEASURES:

1. Primary Outcome: Maximum IVC Diameter
Description: Maximum Inferior Vena Cava diameter in mm
Time Frame: 10 minutes
Measure: Median (Full Range); unit: mm
Groups:
- Cases: Pediatric Patients who were dehydrated
- Controls: Pediatric Patients that were hydrated
Arm/Group | Cases | Controls
Number analyzed (Participants) | 13 | 63
mm | 38 [20 to 84] | 64 [23 to 112]

2. Secondary Outcome: Minimum IVC Diameter
Description: Minimum Inferior Vena Cava Diameter in mm
Time Frame: 10 minutes
Measure: Median (Full Range); unit: mm
Arm/Group | Cases | Controls
Number analyzed (Participants) | 13 | 63
mm | 30 [3 to 57] | 45 [13 to 90]

ADVERSE EVENTS:
Arm/Group | Cases | Controls
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/63
Other Adverse Events (participants affected / at risk) | 0/13 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No